CLINICAL TRIAL: NCT00245219
Title: Understanding Shared Psychobiological Pathways--Project 4. Psychobiological Pathways: Breast Cancer Interventions
Brief Title: Understanding Shared Psychobiological Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael F. Scheier, Professor of Psychology, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 338; P50HL065111 (NIH)
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Health Tracking (control) (No Intervention): Participants assigned to the health-tracking condition received usual care and did not attend any meetings.
- Peer support (Experimental): The peer support group meetings focused on fostering purpose in life by providing participants with opportunities to support and care for one another. Patients completed a weekly diary of critical experiences or current life problems as homework, and were then encouraged to share these experiences in the group meetings. The group facilitator encouraged participants to help one another with these issues, and share how they had dealt with similar problems.
  Interventions: Behavioral: Peer support
- Education (Experimental): The education group meetings focused on providing patients with information about their disease as well as methods to manage their illness and its side effects. Facilitators emphasized the theme of perceived control during all sessions, discussing how participants are in control of their illness experience and can have more control of their lives. A different topic was addressed in each session. Weekly homework assignments asked patients to write down something new they had learned from the session regarding how to take control of their lives. Meeting topics were as follows: Overview of breast cancer, treatment types and side effects, nutrition and diet management, exercise, body image, communication issues, relationships, and sexuality.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — The education group meetings focused on providing patients with information about their disease as well as methods to manage their illness and its side effects. Facilitators emphasized the theme of perceived control during all sessions, discussing how participants are in control of their illness experience and can have more control of their lives. A different topic was addressed in each session. Weekly homework assignments asked patients to write down something new they had learned from the session regarding how to take control of their lives. Meeting topics were as follows: Overview of breast cancer, treatment types and side effects, nutrition and diet management, exercise, body image, communication issues, relationships, and sexuality.
  Arms: Education
Behavioral: Peer support — The peer support group meetings focused on fostering purpose in life by providing participants with opportunities to support and care for one another. Patients completed a weekly diary of critical experiences or current life problems as homework, and were then encouraged to share these experiences in the group meetings. The group facilitator encouraged participants to help one another with these issues, and share how they had dealt with similar problems.
  Arms: Peer support

SUMMARY:
The present study sought to investigate the efficacy of two psychosocial interventions for breast cancer patients, a peer support intervention and an education intervention. The present study also sought to identify mechanisms underlying the benefits of these interventions, and to determine if the efficacy of these interventions is moderated by cancer severity.

DETAILED DESCRIPTION:
BACKGROUND:

The study was a subproject within a Mind-Body Center on Understanding Shared Psychobiological Pathways. The Center was in response to a Request for Applications issued by the Office of the Director, NIH. Dr. Scheier was the Co-Director of the Center as well as the subproject principal investigator. The major objective of the Center was to to identify, measure, and understand the shared psychological, behavioral, and psychobiological pathways that contributed to the onset of and recovery from diverse physical illnesses, which included infections, arthritis, cancer, and cardiovascular disease.

The subproject studied an important area of psychosocial research in cancer, specially the relative effectiveness of different psychosocial interventions for women with breast cancer, and the mechanisms that underlie the benefits of these interventions.

DESIGN NARRATIVE:

The specific aims of the project were to:

1. implement and evaluate two psychosocial interventions, a peer support intervention and an education intervention, to enhance psychological adjustment and well-being among women with early- vs. late-stage breast cancer
2. determine the psychological, behavioral, and biological mechanisms through which the interventions operate
3. assess whether the two interventions were differentially effective for women with different characteristics, most importantly early- vs. late-stage disease
4. use the baseline data collected prior to the intervention to determine the nature and extent of difficulties faced by early- vs. late-stage breast cancer patients
5. determine how participants in the intervention differed from those who choose to participate.

Participants included 180 patients with early stage (I or II) and 65 patients with late stage (IV) breast cancer. The interventions were conducted in groups of 6-9 women, and groups met once a week for 8 weeks. The education group meetings focused on providing patients with information about their disease as well as methods to manage their illness and its side effects. Facilitators emphasized the theme of perceived control during all sessions, discussing how participants are in control of their illness experience and can have more control of their lives. The peer support group meetings focused on fostering purpose in life by providing participants with opportunities to support and care for one another. Participants were asked to share experiences and problems in group meetings and the group facilitator encouraged participants to help one another with these issues, and share how they had dealt with similar problems. Participants in the control condition received care as usual, and did not attend any group meetings.

Hypothesized predictors, mediators, and relevant outcome measures were assessed prior to the intervention. Mediators and outcomes were then reassessed, 2-weeks after intervention completion and 6-months later.

ELIGIBILITY:
Eligible participants were:

1. English speaking women,
2. 25 years of age or older,
3. Living within a 60 mile radius of Pittsburgh, Pennsylvania,
4. either: a first time diagnosis of stage I or II breast cancer or if they had received an initial diagnosis of stage IV cancer or a distant recurrence of breast cancer,
5. Patients with early stage cancer must have been diagnosed within the past 6 months,
6. There was no window for enrollment for patients with late stage cancer.

Ages: 26 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 1999-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scheier, Principal Investigator — Carnegie Mellon University

REFERENCES:
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from local oncologists' offices. We contacted 915 eligible patients, of whom 245 provided informed consent and were randomized to an intervention group. The most frequently reported reasons for refusal were unwillingness/inability to drive to group meeting site (37.2%) and being too busy (29.4%).
Period: Overall Study
Arm/Group | Health Tracking (Control) | Peer Support | Education
Started | 91 | 94 | 60
Completed | 85 | 88 | 58
Not Completed | 6 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Tracking (Control) | Peer Support | Education | Total
Number analyzed (Participants) | 91 | 94 | 60 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.26 (9.56) | 51.40 (10.19) | 49.68 (8.64) | 50.96 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 94 | 60 | 245
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White, Caucasian | 84 | 80 | 56 | 220
  Black, African-American | 6 | 12 | 4 | 22
  Other | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mental Health (as Measured With the SF-36) at Baseline, Time 2 (2 Weeks Post-intervention) and Time 3 (6 Months Post-intervention)
Description: The Mental Health Component Scale of the Medical Outcomes Study Short Form 36(SF-36) consists of a norm-based weighted average of the following subscales: Vitality, Social Functioning, Role Limitations due to Emotional Problems and Mental health. In the present study, scores ranged from a maximum of 72 (high levels of mental health) to a minimum of 12 (low levels of mental health).
Time Frame: Baseline, Time 2 (2 weeks post-intervention) and Time 3 (6 months post-intervention)
Population: The intention-to-treat principle was followed, all participants were included in the analyses regardless of number of meetings attended.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Tracking (Control) | Peer Support | Education
Number analyzed (Participants) | 85 | 62 | 46
units on a scale
  Baseline | 46.55 (11.61) | 47.63 (11.25) | 47.12 (11.27)
  Time 2 | 47.03 (10.40) | 49.25 (10.64) | 50.67 (11.22)
  Time 3 | 50.28 (9.88) | 50.03 (11.18) | 48.02 (13.10)
Statistical Analysis 1: Comparison: Health Tracking (Control) vs Peer Support; The comparison between the peer support condition and the control condition at Time 2. The full regression model included 2 dummy coded variables, 1 contrasting the education and control condition, and 1 contrasting the peer support and control condition. The baseline measure of the outcome variable was included, in order to examine changes in the outcomes over time. This model tested the main effects of the conditions among patients with early stage cancer, late stage patients were excluded; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Health Tracking (Control) vs Education; The comparison between the education condition and the control condition at Time 2. The full regression model included 2 dummy coded variables, 1 contrasting the education and control condition, and 1 contrasting the peer support and control condition. The baseline measure of the outcome variable was included, in order to examine changes in the outcomes over time. This model tested the main effects of the conditions among patients with early stage cancer, late stage patients were excluded; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 3: Comparison: Health Tracking (Control) vs Peer Support; The comparison between the peer support condition and the control condition at Time 3. The full regression model included 2 dummy coded variables, 1 contrasting the education and control condition, and 1 contrasting the peer support and control condition. The baseline measure of the outcome variable was included, in order to examine changes in the outcomes over time. This model tested the main effects of the conditions among patients with early stage cancer, late stage patients were excluded; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 4: Comparison: Health Tracking (Control) vs Education; The comparison between the education condition and the control condition at Time 3. The full regression model included 2 dummy coded variables, 1 contrasting the education and control condition, and 1 contrasting the peer support and control condition. The baseline measure of the outcome variable was included, in order to examine changes in the outcomes over time. This model tested the main effects of the conditions among patients with early stage cancer, late stage patients were excluded; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 5: Comparison: Health Tracking (Control) vs Peer Support; The comparison between the peer support condition and control condition at Time 2, among both late and early stage patients. The full regression model consisted of 3 steps: The 1st step contained the baseline measure of the dependent variable. The 2nd step contained two dummy coded variables contrasting each condition with control. The 3rd step contained the interaction between the peer support condition and cancer stage. Patients in the education condition were excluded from this analysis; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 6: Comparison: Health Tracking (Control) vs Peer Support; The comparison between the peer support condition and control condition at Time 3, among both late and early stage patients. The full regression model consisted of 3 steps: The 1st step contained the baseline measure of the dependent variable. The 2nd step contained two dummy coded variables contrasting each condition with control. The 3rd step contained the interaction between the peer support condition and cancer stage. Patients in the education condition were excluded from this analysis; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 7: Comparison: Health Tracking (Control) vs Peer Support; The interaction between the peer support condition and cancer stage at Time 2. The full regression model consisted of 3 steps: The 1st step contained the baseline measure of the dependent variable. The 2nd step contained two dummy coded variables contrasting each condition with control. The 3rd step contained the interaction between the peer support condition and cancer stage. Patients in the education condition were excluded from this analysis; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 8: Comparison: Health Tracking (Control) vs Peer Support; The interaction between the peer support condition and cancer stage at Time 3. The full regression model consisted of 3 steps: The 1st step contained the baseline measure of the dependent variable. The 2nd step contained two dummy coded variables contrasting each condition with control. The 3rd step contained the interaction between the peer support condition and cancer stage. Patients in the education condition were excluded from this analysis; Test type: Superiority or Other; p > 0.05, Regression, Linear

2. Primary Outcome: Perceived Physical Health (as Measured With the SF36) at Baseline, Time 2 (2 Weeks Post-intervention) and Time 3 (6 Months Post-intervention)
Description: The Perceived Physical Health Component scale of the Medical Outcomes Study Short Form 36(SF-36) consists of a norm-based weighted average of the following subscales: Physical Functioning, Bodily Pain, Role Limitations due to Physical Problems and General Health. In the present study, scores ranged from a maximum of 70 (high levels of perceived health) to a minimum of 12 (low levels of perceived health).
Time Frame: Baseline, Time 2 (2 weeks post-intervention) and Time 3 (6 months post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Tracking (Control) | Peer Support | Education
Number analyzed (Participants) | 85 | 62 | 46
units on a scale
  Baseline | 42.43 (9.39) | 44.40 (8.93) | 47.62 (8.81)
  Time 2 | 43.46 (11.23) | 46.49 (11.02) | 50.47 (7.56)
  Time 3 | 46.02 (11.53) | 47.36 (11.43) | 51.96 (8.96)
Statistical Analysis 1: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Health Tracking (Control) vs Education; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 3: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 4: Comparison: Health Tracking (Control) vs Education; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 5: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 6: Comparison: Health Tracking (Control) vs Peer Support; The interaction between the peer support condition and breast cancer stage at Time 2. The full regression model consisted of 3 steps: The 1st step contained the baseline measure of the dependent variable. The 2nd step contained two dummy coded variables contrasting each condition with control. The 3rd step contained the interaction between the peer support condition and cancer stage. Patients in the education condition were excluded from this analysis; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 7: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 8: Comparison: Health Tracking (Control) vs Peer Support; The interaction between the peer support condition and breast cancer stage at Time 3. The full regression model consisted of 3 steps: The 1st step contained the baseline measure of the dependent variable. The 2nd step contained two dummy coded variables contrasting each condition with control. The 3rd step contained the interaction between the peer support condition and cancer stage. Patients in the education condition were excluded from this analysis; Test type: Superiority or Other; p > 0.05, Regression, Linear

3. Primary Outcome: Depressive Symptoms (as Measured With the CES-D) at Baseline, Time 2 (2 Weeks Post-intervention) and Time 3 (6 Months Post-intervention)
Description: Scores for the shortened form of the Center for Epidemiologic Studies Depression scale(CES-D) ranged from 0 (no depressive symptoms) to 29 (high levels of depressives symptoms) in the present sample. For the sake of analyses, CES-D scores were dichotomized (cutoff score of 8), because scores exhibited marked positive skew in the present sample.
Time Frame: Baseline, Time 2 (2 Weeks post-intervention) and Time 3 (6 months post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Tracking (Control) | Peer Support | Education
Number analyzed (Participants) | 85 | 62 | 46
units on a scale
  Baseline | 7.78 (6.05) | 6.14 (5.15) | 7.37 (6.61)
  Time 2 | 8.53 (5.80) | 6.75 (5.89) | 6.37 (6.02)
  Time 3 | 6.94 (5.45) | 6.19 (5.92) | 6.60 (6.55)
Statistical Analysis 1: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Regression, Logistic
Statistical Analysis 2: Comparison: Health Tracking (Control) vs Education; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p > 0.05, Regression, Logistic
Statistical Analysis 3: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p > 0.05, Regression, Logistic
Statistical Analysis 4: Comparison: Health Tracking (Control) vs Education; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p > 0.05, Regression, Logistic
Statistical Analysis 5: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p > 0.05, Regression, Logistic
Statistical Analysis 6: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p > 0.05, Regression, Logistic
Statistical Analysis 7: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p > 0.05, Regression, Logistic
Statistical Analysis 8: Comparison: Health Tracking (Control) vs Peer Support; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; p > 0.05, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | Health Tracking (Control) | Peer Support | Education
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/94 | 0/60
Other Adverse Events (participants affected / at risk) | 0/91 | 0/94 | 0/60

LIMITATIONS AND CAVEATS:
The study was originally planned as a 2(early stage, late stage) X 3(education intervention, peer support intervention, control condition) design; however, the education condition for the late stage cancer group was dropped, due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No